CLINICAL TRIAL: NCT01106911
Title: Assessment of Digital Breast Tomosynthesis (DBT) in the Screening Environment: a Prospective Study
Brief Title: Assessment of Digital Breast Tomosynthesis (DBT) in the Screening Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jules Sumkin, Chief of Women's Imaging, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO09060334
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Breast Abnormalities
Keywords: digital breast tomosynthesis; baseline screening mammography; recall rates
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: tomosynthesis and screening mammography — All eligible subjects will undergo both full field digital mammography and digital breast tomosynthesis.
  Other Names: digital breast tomosynthesis

SUMMARY:
The objective of this study is to demonstrate that digital breast tomosynthesis (DBT) in combination with full field digital mammography (FFDM) has the potential to reduce significantly baseline screening recall rates without a loss in the detection of cancers. The primary hypothesis of the study is that DBT in combination with FFDM will reduce baseline screening mammography recall rates in negative examinations by at least 20%.

DETAILED DESCRIPTION:
The FFDM images and the FFDM images with the DBT images will be interpreted independently by two experienced radiologists under standard clinical screening procedures. Recommended recall rates will be assessed and compared as a result of each of the two interpretations.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 34 and 56.
* Women presenting for their baseline screening mammography examination

Exclusion Criteria:

* Women with a palpable finding(s) via a Breast Self Examination (BSE) or Clinical Breast Examination (CBE).
* Women who may be or are pregnant by self report
* Women older than 55 years of age or younger than 35.
* Women with known fatty breast tissue
* Males and children
* Women who are unable to understand or execute written informed consent

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1080 (Actual)
Dates: Start 2010-05; Primary Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jules H Sumkin, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were consented, screened and enrolled at one site, a medical hospital specializing in women's health. The period of recruitment was from May, 2010 to September, 2014.
Pre-assignment Details: Three subjects were deemed ineligible. Two subjects were withdrawn by the PI after beginning research procedures.
Groups:
- Digital Breast Tomosynthesis (DBT): Consented and eligible women undergoing baseline screening mammography received DBT
Period: Overall Study
Arm/Group | Digital Breast Tomosynthesis (DBT)
Started | 1085
Completed | 1080
Not Completed | 5
Not completed — Physician Decision | 2
Not completed — deemed ineligible after screening | 3

BASELINE CHARACTERISTICS:
Population: Participants who completed research procedures
Arm/Group | Digital Breast Tomosynthesis (DBT)
Number analyzed (Participants) | 1080
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.03 (3.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1080
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 1054
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 35
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 278
  White | 751
  More than one race | 0
  Unknown or Not Reported | 16
Region of Enrollment [Number; unit: participants]
  United States | 1080

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Cancer Who Were Recalled
Description: Recall rates of digital breast tomosynthesis and full field digital mammography in younger women undergoing their initial screening mammogram will be assessed and compared.
Time Frame: upon recruitment/enrollment phase completion
Population: Includes only participants who were not diagnosed as having a breast malignancy.
Measure: Number; unit: participants
Arm/Group | Digital Breast Tomosynthesis (DBT)
Number analyzed (Participants) | 1074
participants | 274

ADVERSE EVENTS:
Time Frame: 1 day
Description: The technologist performing DBT documented the skin condition of the participant and reported if any acute injury occurred during the exam.
Arm/Group | Digital Breast Tomosynthesis (DBT)
Serious Adverse Events (participants affected / at risk) | 0/1080
Other Adverse Events (participants affected / at risk) | 0/1080

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No